CLINICAL TRIAL: NCT05433428
Title: Metabolomic Profile in Tear Film Samples of Patients With or Without Dry Eye Syndrome Before and After Cataract Surgery.
Brief Title: Metabolomic Profile in Dry Eye Syndrome Patients.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ifocus Oyeklinikk (Network)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 140664
Record Dates: First submitted 2020-08-10; First posted 2022-06-27 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Dry Eye Syndromes; Cataract
Keywords: Metabolomics; Dry Eye Syndrome; Cataract surgery
MeSH Terms: conditions — Dry Eye Syndromes; Cataract | interventions — Lubricant Eye Drops; Preservatives, Pharmaceutical

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cataract patients with dry eye - standard treatment (Experimental): Standard pre and postop medication, preservative eye drops.
  Interventions: Drug: Preservative
- Cataract patients with dry eye - intensive treatment (Other): More prolonged use of lubricant eye drops as well as the use of preservative free eye drops.
  Interventions: Drug: Lubricant Eye Drops; Drug: Preservative Free
- Cataract patients without dry eye disease / control group (Other): Standard pre and postop medication, control group.
  Interventions: Drug: Preservative

INTERVENTIONS:
Drug: Lubricant Eye Drops — Prolonged use of lubricant eye drops pre and post-op.
  Arms: Cataract patients with dry eye - intensive treatment
Drug: Preservative Free — Preservative free eye drops
  Arms: Cataract patients with dry eye - intensive treatment
Drug: Preservative — Eyedrops with preservatives
  Arms: Cataract patients with dry eye - standard treatment; Cataract patients without dry eye disease / control group

SUMMARY:
The primary objective is to determine possible implications of deviant tear film quality for optimal refractive precision in patients scheduled for cataract surgery.

The study consist of three separate arms where cataract patients will be separated in to Dry Eye Disease (DED) positive and negative groups. The DED positive group will be further subdivided into two different treatment groups (with focus on prolonged use of lubricant and preservative free eye drops). Tear film samples will be taken before treatment, after treatment and after surgical treatment and compared.

DETAILED DESCRIPTION:
The participants will be randomized to either standard pre- and postoperative treatment protocol - hereby called the standard protocol - or a pre- and postoperative protocol where intensive dry eye treatment is implemented - hereby called the intensive dry eye treatment protocol. The intensive dry eye treatment protocol differs from the standard protocol in the use of preservative free eye drops and the use of topical steroids prior to surgery.

The standard treatment protocol is:

Before surgery:

* Nevanac 3 mg /mL
* Spersadex 1mg/ml three days before surgery.

After surgery:

Nevanac 3 mg /mL five days after surgery. Spersadex 1 mg/ml 20 days after surgery

The intensive dry eye treatment protocol is:

Before surgery:

Lubricants (Thealoz Duo) for four weeks. Preservative free dexamethasone 0.1% (Monopex) drops for one week Preservative free Diklofenak 1mg/mL drops (Voltaren minims) four times a day from three days before surgery.

After surgery:

Lubricants (Thealoz Duo) for three weeks. Preservative free dexamethasone 0.1% (Monopex) drops for three weeks. Preservative free Diklofenak 1mg/mL drops (Voltaren minims) for five days after surgery.

Biometry will be performed prior to and after the preoperative treatment, 6 weeks after surgery.

The variability in biometry measurements will be assessed for the standard protocol group versus the intensive dry eye protocol group. In addition, the average difference in estimated refraction and the actual refractive outcome (deltaR) will be calculated for both groups.

Differences in tear film instability before and after preoperative treatment, 6 weeks after surgery will be investigated.

Other variables to be investigated:

Average corneal curvature (K) Anterior corneal curvature Corneal astigmatism Mean spherical equivalent Dioptric keratometric power (estimated Intraocular lens (IOL) power) Best corrected visual acuity Tearlab osmolarity Non-invasive break up time(NIBUT) Tear meniscus height Bulbar redness grade Tear film lipid layer thickness (Lipiview) Ocular scatter analysis (HD analyzer) Cochet-Bonnet esthesiometry Ocular surface staining(OSS) Schirmers I test (without anesthetics) Meibum expressibility Meibum quality Meibomian gland dropout (meibography) Lid margin irregularities (yes/no) Tarsal conjunctival follicles/papillae (yes/no) Ocular surface disease index(OSDI) Dry Eye Quality of life questionnaire-5 (DEQ-5) Standard Patient Evaluation of Eye Dryness II (SPEED II)

ELIGIBILITY:
Inclusion Criteria:

* Indication for cataract surgery
* Signed informed consent
* no rheumatological or other systemic disease that involve the corneal surface
* a good ocular health with no pathology that compromises visual acuity (except cataract).

Exclusion Criteria:

* Manifest corneal disease or scarring
* Lid deformities
* Corneal ectasia
* Rheumatoid diseases or other systemic diseases that involve the corneal surface,
* Recent ocular surgery
* Previous refractive procedures
* Diabetic retinopathy
* Subjects who have an acute or chronic disease or illness that would confound the results of this investigation (e.g., immunocompromised, connective tissue disease, clinically significant atopic disease, diabetes, and any other such disease or illness)
* Pregnancy.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2020-08-03 (Actual); Primary Completion 2023-01-10 (Estimated); Study Completion 2023-05-23 (Estimated)

PRIMARY OUTCOMES:
Metabolomic and lipodomic profile | 6 weeks
  The metabolomic and lipodomic profiles of the tears in each group will be measured. Relevant metabolic/lipid results will be reported.

SECONDARY OUTCOMES:
Spherical equivalent refraction | 6 weeks
  Spherical equivalent refraction in diopters.
Refractive cylinder | 6 weeks
  Refractive cylinder in diopters.

CONTACTS AND LOCATIONS:
Overall Officials: Morten Gundersen, MD, Principal Investigator — IFocus Øyeklinikk AS
Locations (1):
- Ifocus øyeklinikk, Haugesund, Norway

IPD SHARING:
Plan to Share IPD: No